CLINICAL TRIAL: NCT03747497
Title: A Phase 2, Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Contezolid Acefosamil Compared to Linezolid Administered Intravenously and Orally to Adult Subjects With Acute Bacterial Skin and Skin Structure Infection
Brief Title: Contezolid Acefosamil Versus Linezolid for the Treatment of Acute Bacterial Skin and Skin Structure Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MicuRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRX4-201
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Results first posted 2021-04-30 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Skin Diseases, Bacterial; Gram-Positive Bacterial Infections
Keywords: ABSSSI; Acute bacterial skin and skin structure infection
MeSH Terms: conditions — Skin Diseases, Bacterial; Gram-Positive Bacterial Infections | interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- contezolid acefosamil (Experimental): contezolid acefosamil 1500 mg IV x 1 dose, followed by 1000 mg IV q12h for at least 3 total IV doses, followed by 1300 mg PO q12h for 10 to 14 days
  Interventions: Drug: contezolid acefosamil
- linezolid (Active Comparator): linezolid 600 mg IV q12h for at least 3 total IV doses, followed by 600 mg PO q12h for 10 to 14 days
  Interventions: Drug: linezolid 600 mg

INTERVENTIONS:
Drug: contezolid acefosamil — IV and oral contezolid acefosamil given twice a day for 10 to 14 days
  Arms: contezolid acefosamil
Drug: linezolid 600 mg — IV and oral linezolid given twice a day for 10 to 14 days
  Other Names: Zyvox
  Arms: linezolid

SUMMARY:
The purpose of this study is to determine whether contezolid acefosamil is as safe and effective as linezolid in the treatment of adult patients with acute bacterial skin and skin structure infections

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic signs of infection diagnosed with acute bacterial skin and skin structure infection (ABSSSI)
* Diagnosed with cellulitis/erysipelas, major cutaneous abscess, or wound infections

Exclusion Criteria:

* Uncomplicated skin infections
* Severe sepsis or septic shock
* ABSSSI solely due to Gram-negative pathogens
* Prior systemic antibiotics within 96 hours of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - MicuRx Site #106, Chula Vista, California
  - MicuRx Site #103, La Mesa, California
  - MicuRx Site #102, Long Beach, California
  - MicuRx Site #104, Stockton, California
  - MicuRx Site #107, Butte, Montana
  - MicuRx Site #105, Las Vegas, Nevada
  - MicuRx Site #108, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 196 subjects were randomized
Groups:
- Contezolid Acefosamil: Contezolid acefosamil 1500 IV x 1 dose, followed by 1000 mg IV q12h, for at least 3 total IV doses, followed by 1300 mg PO q12h
- Linezolid: Linezolid 600 mg IV q12h, for at least 3 total IV doses, followed by 600 mg PO q12h
Period: Overall Study
Arm/Group | Contezolid Acefosamil | Linezolid
Started | 131 | 65
Completed | 106 | 55
Not Completed | 25 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contezolid Acefosamil | Linezolid | Total
Number analyzed (Participants) | 131 | 65 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (11.87) | 43.7 (10.94) | 44.5 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 18 | 70
  Male | 79 | 47 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 28 | 79
  Not Hispanic or Latino | 80 | 37 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 109 | 58 | 167
  Black or African American | 8 | 4 | 12
  Asian | 2 | 1 | 3
  American Indian or Alaska Native | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Other | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response at the Early Assessment Visit (ITT Population)
Description: Early clinical response assessment based on the electronic case report form (eCRF) data at Early Assessment (48-72 hours after start of study drug) where a successful response (i.e., "responder") was defined as a reduction in primary ABSSSI lesion size ≥20% compared to baseline, and the subject did not receive a non-protocol specified systemic antibacterial agent with activity against Gram-positive organisms for the treatment of ABSSSI and did not die of any cause up to Early Assessment.
Time Frame: 48 to 72 hours after the start of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Contezolid Acefosamil | Linezolid
Number analyzed (Participants) | 131 | 65
Participants
  Responder | 102 | 51
  Non-Responder | 3 | 6
  Indeterminate | 26 | 8
Statistical Analysis 1: Comparison: Contezolid Acefosamil vs Linezolid; Test type: Other; Median Difference (Net) = -0.6, 95% CI 2-sided [-14.0 to 2.8]

ADVERSE EVENTS:
Time Frame: 28 Days
Description: The ITT Population (N=131) consists of all randomized subjects regardless of whether or not the subject received study drug. The Safety Population consists of all randomized subjects who received any amount of study drug, and included 123 subjects in the contezolid acefosamil group and 64 subjects (98.5%) in the linezolid group. All safety analyses were conducted in this population and were analyzed by the treatment the subject actually received.
Arm/Group | Contezolid Acefosamil | Linezolid
All-Cause Mortality (participants affected / at risk) | 1/123 | 1/64
Serious Adverse Events (participants affected / at risk) | 3/123 | 1/64
Other Adverse Events (participants affected / at risk) | 55/123 | 27/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Contezolid Acefosamil (N=123) | Linezolid (N=64)
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Contezolid Acefosamil (N=123) | Linezolid (N=64)
Nausea (Gastrointestinal disorders) | 18 | 5
Vomiting (Gastrointestinal disorders) | 9 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Cellulitis (Infections and infestations) | 9 | 7
Abscess (Infections and infestations) | 6 | 2
Wound infection (Infections and infestations) | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 0
Injection site extravasation (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 1 | 2
Headache (Nervous system disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT03747497/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT03747497/SAP_001.pdf